CLINICAL TRIAL: NCT02921464
Title: Florida Cardiovascular Quality Network
Acronym: FCQN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Florida Cardiovascular Quality Network (Other)
Responsible Party: Principal Investigator, William David, MD, FACC, Director, Florida Cardiovascular Quality Network, Florida Cardiovascular Quality Network
Other Study IDs: 201600631
Record Dates: First submitted 2016-08-08; First posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Stable Ischemic Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Group A - without known pre-existing SIHD
  Interventions: Other: none - registry clinic followup only
- Group B: Group B - with known pre-existing SIHD.
  Interventions: Other: none - registry clinic followup only

INTERVENTIONS:
Other: none - registry clinic followup only

SUMMARY:
Florida Cardiovascular Quality Network Application of Clinical Decision Support Software Tools at the Point of Care in Patients with Stable Ischemic Heart Disease - a Quality Outcomes Registry

DETAILED DESCRIPTION:
The Florida Cardiovascular Quality Network (FCQN) is a quality outcomes registry. In a diverse group of clinical sites in Florida, a large number of patients with known or possible stable ischemic cardiovascular disease (SIHD) referred for cardiovascular stress test will be enrolled in this quality demonstration registry. This registry is based on the hypothesis that evidence-based clinical guidelines and appropriate use criteria (AUC), when provided at the site and time of care (point of care), may improve physician clinical decisions and, thus, the overall quality and value of care for individual patients and populations. Specifically, this study registry will utilize multiple proven software tools at the point of care: (1) Seattle Angina Questionnaire (SAQ) as the method of measurement of patient angina symptoms; (2) FOCUS, American College of Cardiology (ACC) software to provide clinical decision support (CDS) as the primary method of determination of AUC in patients with a clinical indication for a cardiovascular stress test; (3) CATH/PCI, ACC / National Cardiovascular Data Registry (NCDR) to provide clinical decision support as the primary method of determination of AUC in the cardiac catheterization laboratory; (4) PINNACLE, ACC/NCDR clinical registry to provide an extensive database of clinical quality metrics; and (5) ACC CARDIOSMART software modules as the primary patient education tool for effective risk factor modification. The application of these clinically proven software tools, all applied at the point of patient care, may assist physician compliance with ACC guideline based AUC and may directly result in an increase in SIHD patients treated with guideline directed medical treatment as well as guideline directed interventional treatment. It is anticipated that this increased compliance with ACC guidelines and AUC may directly correlate with improved patient clinical outcomes.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patient presents for evaluation of SIHD and meets patient eligibility criteria as defined as SIHD Group A or SIHD Group B patient.
2. Patient is over 21 years of age
3. Patient is a stable clinic patient with the intention to continue in continuous medical care for the duration of the registry.

EXCLUSION CRITERIA:

1. Patient is diagnosed with acute coronary syndrome (unstable angina, myocardial infarction -either non-STEMI or STEMI)
2. Patient has a concomitant medical illness that may limit survival to less than 1 year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group A patients will be identified by no established SIHD, but presenting with symptoms consistent with myocardial ischemia; Group B patients will be idenitified by Established SIHD and symptoms of myocardial ischemia. All patients will have: (1) Indications for functional stress testing. All functional stress tests will be designed to provoke cardiac ischemia by using exercise or pharmacological stress agents; (2) Multiple (>3) cardiac risk factors including male gender, age > 50 years old, diabetes mellitus, hypertension, hyperlipidemia, nicotine exposure, and/or family history of cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Angina Classification | 1 year
  Angina Classification derived from Seattle Angina Questionaire (SAQ)
Appropriate Use Criteria (AUC) for Stress Test | 1 year
  AUC derived from FOCUS clinical decision support software
Appropriate Use Criteria (AUC) for Coronary Intervention | 1 year
  AUC derived from CATH/PCI data
Fractional Flow Reserve (FFR) | 1 year
  FFR derived from CATH/PCI data

SECONDARY OUTCOMES:
Composite Adverse Cardiac Events - Death, Myocardial Infarction, Hospitalization for Acute Coronary Syndrome - correlate with Angina Classification, SAQ, and AUC for Stress Testing | 1 year
  Adverse Cardiac Events derived from case report form and PINNACLE database
Composite Adverse Cardiac Events - Death, Myocardial Infarction, Hospitalization for Acute Coronary Syndrome - correlate with Coronary Intervention AUC and FFR | 1 year
  Adverse Cardiac Events derived from case report form and PINNACLE database

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Center, Lake Mary, Florida, United States

IPD SHARING:
Plan to Share IPD: No